CLINICAL TRIAL: NCT07257354
Title: Reducing Examination Anxiety Through Emotional Freedom Techniques: A Randomized Controlled Trial Among Somali Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSTH/9570
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Emotional Freedom Techniques
Keywords: Emotional Freedom Techniques; Stress coping; Exam anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFT Group (Experimental): Participants in the intervention group received two 45-55 minute EFT sessions one week before the exam.
  Interventions: Other: Emotional Freedom Technique
- Breath Group (Experimental): Participants in the comparison group received two sessions of 15-20 minutes of breathing exercises one week before the exam.
  Interventions: Other: Breath Group

INTERVENTIONS:
Other: Emotional Freedom Technique — The EFT group received two 45-55 minute EFT sessions one week before the exams.
  Arms: EFT Group
Other: Breath Group — The breathing group received two sessions of 15-20 breathing exercises a week before the exams.
  Arms: Breath Group

SUMMARY:
This study aims to determine the effects of the Emotional Freedom Technique applied before exams on coping with stress and anxiety.

DETAILED DESCRIPTION:
This experimental randomized controlled trial assigned participants to two groups: the EFT Group (n=31) and the Breathing Group (n=31). Each group received two intervention sessions, held one week apart, prior to the midterm exams. Final assessments were conducted one week after the exams. Data collection tools included the Visual Analog Scale for Anxiety to measure anxiety levels, and the Coping Styles with Stress Scale.

ELIGIBILITY:
Inclusion Criteria:

* Turkish proficiency, willingness to participate in the study voluntarily

Exclusion Criteria:

* The student has coordination and language problems, any diagnosed psychiatric disorder or epilepsy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | 10 minütes
  Anxiety levels were assessed using the Visual Analog Scale. Students were asked to indicate their anxiety levels on a 10-cm-long horizontal line. The line begins with a 0 and ends with a 10. A 10 indicates extreme anxiety, while a 0 indicates no anxiety. The VAS scale is frequently used to assess anxiety severity.
Stress Coping Styles | 10 minütes
  The Styles of Coping Scale (SCSS) was used to measure stress coping styles. The scale is a 4-point Likert-type scale, with participants selecting the appropriate option from "not at all appropriate" to "very appropriate." The scale consists of 30 questions and 5 subscales. These subscales are: self-confident approach, optimistic approach, helpless approach, submissive approach, and seeking social support factor. Higher scores on each subscale indicate that the approach in that subscale is used more frequently to cope with stress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)